CLINICAL TRIAL: NCT00591305
Title: Voice Preserving Therapy of Laryngeal Papilloma In Children
Brief Title: New Therapy of Laryngeal Papilloma In Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient resource for recruitment
Sponsor: Boston University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Zhi Wang, Professor and Director, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RDC-008287A; 5R01DC008287 (NIH)
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Papilloma
Keywords: papilloma; PDL; diindolylmethane; recurrence
MeSH Terms: conditions — Papilloma; Recurrence | interventions — 3,3'-diindolylmethane; Lasers, Dye

STUDY DESIGN:
Intervention Model Description: laser only vs laser+ a dietary agent (DIM)
Who Masked: Participant
Masking Description: treatment to be selected based on a randomized number table, blinded to participants
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDL+DIM pill (Experimental): once-time 585 nm pulsed dye laser (PDL) treatment on the lesions, immediately followed by 3-month oral taking diindolylmethane (DIM, at 1.2-1.75mg/kg/day), in 15 subjects
  Interventions: Dietary Supplement: diindolylmethane (DIM); Device: 585 nm pulsed dye laser
- PDL+placebo pill (Placebo Comparator): once-time PDL treatment on the lesions, then followed by 3-month oral taking DIM placebo, in other 15 subjects
  Interventions: Device: 585 nm pulsed dye laser

INTERVENTIONS:
Dietary Supplement: diindolylmethane (DIM) — 3-month DIM
  Arms: PDL+DIM pill
Device: 585 nm pulsed dye laser — once-time PDL

SUMMARY:
This study will determine efficacy of a new and combined treatment of laryngeal recurrent respiratory papillomatosis (RRP), by using a 585 nm pulsed dye laser (PDL) and a dietary supplement, diindolylmethane (DIM). We will compare this new treatment with PDL-only, in a total of 30 children (15 of each treatment), to determine whether this combined treatment would be effective and safe in preventing the RRP recurrence. This is the first study to combine PDL technique with DIM, to develop a new, voice-preserving and long-term effective method of managing laryngeal RRP in children.

DETAILED DESCRIPTION:
Previous studies have demonstrated that PDL can be used to remove lesions on the vocal cords and elsewhere in the throat causing less damage to surface tissues than other commonly used lasers. In our proposed clinical study, we seek to compare treatment efficacy for RRP by combining PDL with DIM, versus PDL-only treatment, in a total of 30 children with laryngeal papilloma. We will determine whether this combined treatment would be effective and safe in preventing or delaying the RRP recurrence while preserving voice quality. 30 children will be divided randomly into two treatment groups, 15 in each. The experimental group will receive one-time PDL treatment, followed by 3-month oral administration of DIM and an additional 12 months with no treatment. The other group will be treated with PDL-only, as a control, and take a placebo pill for 3 months. All of the patients will be followed for a total of 15 months. We will compare lesion recurrence and laboratory tests between the two groups, to determine efficacy and safety of the new treatment. This is the first study to combine new PDL laser technique with DIM, to develop a new, voice-preserving and long-term effective method of managing laryngeal RRP in children.

ELIGIBILITY:
Inclusion Criteria:

1. 10 to 21 years of age
2. laryngeal papillomas requiring surgical treatment
3. willingness to participate in the study
4. a signed informed consent form by guardian or parent

Exclusion Criteria:

1. age less than 10 year old, or older than 21 year
2. guardian or parent does not understand or can not sign the consent form
3. malignant diseases such as laryngeal cancer
4. history of being hypersensitive to cabbage or other cruciferous vegetables
5. pregnancy

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Wang, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no such meaningful data available due to insufficient recruitment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 month follow up study
Pre-assignment Details: There was only one participant due to difficulty in recruitment which resulted in early termination of the trial.
Period: Overall Study
Arm/Group | PDL+DIM Pill | PDL+Placebo Pill
Started | 1 | 0
1st Follow-up in 2 Wks After Surgery | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There was only one participant due to difficulty in recruitment which resulted in early termination of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | PDL+DIM Pill | PDL+Placebo Pill | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases With Recurrence of Laryngeal Papilloma in 5 Months
Description: vocal lesion size and area after 5 month with surgery visible lesion found in >50% of the treated tissue area, after surgery
Time Frame: Recurrence of pailloma at 5 months
Population: participants received at least one of two interventions
Measure: Number; unit: case
Groups:
- Intervention: laser+dietary DIM
- Placebo: laser only without DIM
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 1 | 0
case | 1 |

2. Secondary Outcome: Estradiol Level in Blood Pre Treatment
Description: determine side-effect by comparing Estradiol level in blood before and after treatment
Time Frame: Before treatment at baseline
Population: failure for any meaningful analysis as only 1 participant in this study
Measure: Number; unit: pg/ml
Groups:
- Intervention: laser+diatary DIM
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 1 | 0
pg/ml | 20 |

3. Secondary Outcome: Estradiol Level in Blood Post Treatment
Description: determine side-effect by comparing Estradiol level in blood before and after treatment
Time Frame: 5 month
Population: failure for any meaningful analysis as only 1 participant in this study
Measure: Number; unit: pg/ml
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 1 | 0
pg/ml | 29 |

ADVERSE EVENTS:
Time Frame: 3 months after surgery
Groups:
- PDL+Placebo Pill: once-time PDL treatment by PDL on the lesions, then followed by 3-month oral taking DIM placebo, in other 15 subjects
Arm/Group | PDL+DIM Pill | PDL+Placebo Pill
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
There was only one participant due to difficulty in recruitment which resulted in early termination of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No